CLINICAL TRIAL: NCT00507481
Title: Evaluation of Risk Factors of Sleep Quality in Critically Ill Patients
Brief Title: Evaluation of Risk Factors of Sleep Quality in Intensive Care Unit
Status: Completed | Type: Observational
Sponsor: University of Turin, Italy (Other)
Responsible Party: Trompeo Anna Chiara, University of Turin
Other Study IDs: 4627
Record Dates: First submitted 2007-07-24; First posted 2007-07-26 (Estimated); Last update posted 2008-06-04 (Estimated); Status verified 2008-06

CONDITIONS: Sleep Disorders; Delirium
Keywords: Sleep; ICU; Delirium; Post surgical ventilated patients; ICU patients
MeSH Terms: conditions — Sleep Wake Disorders; Delirium

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study was to investigate the relationship between sleep disturbances and delirium in surgical ICU patients. The study set up to test the hypothesis that the occurrence of delirium is associated to the alteration of sleep quality and quantity observed in the critically ill patients.

DETAILED DESCRIPTION:
Sleep disorders are an important clinical entity affecting outcome in respiratory, cardiovascular, metabolic and psychiatric disorders and exacting a potentially significant toll on patients at both a personal and socio-economic level.Delirium is a common organ dysfunction in the critically ill patients characterized by an acute onset of impaired cognitive function [REF] associated with prolonged ICU and hospital stay, nosocomial pneumonia, and death.

ELIGIBILITY:
Inclusion Criteria:

* Adult, postsurgical patients who needed mechanical ventilation for more than 48 hr admitted to the general ICU

Exclusion Criteria:

* Defined a priori
* Were history of chronic dementia, psychosis, mental retardation, stroke syndrome or other primary neurologic disease
* Patient refusal to participate
* Alcohol and drug abuse.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU postsurgical patients who needed mechanical ventilation for more than 48 hr admitted to the general ICU
Sampling Method: Probability Sample
Dates: Start 2006-01; Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marco V Ranieri, Professor, Study Director — University of Turin, Italy
Locations (2):
- Italy (2):
  - Intensive care Unit S.giovanni Battista Hospital, Turin, Turin
  - ICU University S.G.Battista Hospital, Turin